CLINICAL TRIAL: NCT07015905
Title: A Phase 3, Multicenter, Randomized, Open-Label, Sponsor-Blinded, Study to Evaluate REGN7508, A Factor XI Monoclonal Antibody, Versus Apixaban and Enoxaparin for Prophylaxis of Venous Thromboembolism After Elective Total Knee Arthroplasty (ROXI-APEX)
Brief Title: REGN7508 Versus Apixaban and Enoxaparin for Thromboprophylaxis After Total Knee Arthroplasty in Adults
Acronym: ROXI-APEX
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R7508-DVT-24116; 2025-520478-20-00 (EU CTIS Number)
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Venous Thromboembolism (VTE)
Keywords: Unilateral Total Knee Arthroplasty (TKA); Factor XI (FXI)
MeSH Terms: conditions — Venous Thromboembolism | interventions — apixaban; Enoxaparin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- IV REGN7508 (Experimental)
  Interventions: Drug: REGN7508
- IV Placebo, SC REGN7508 (Experimental)
  Interventions: Drug: REGN7508; Drug: Placebo
- IV Placebo, apixaban (Active Comparator)
  Interventions: Drug: Apixaban; Drug: Placebo
- IV Placebo, enoxaparin (Active Comparator)
  Interventions: Drug: Enoxaparin; Drug: Placebo

INTERVENTIONS:
Drug: REGN7508 — Administered per the protocol
  Arms: IV Placebo, SC REGN7508; IV REGN7508
Drug: Apixaban — Administered per the protocol
  Arms: IV Placebo, apixaban
Drug: Enoxaparin — Administered per the protocol
  Other Names: Inhixa
  Arms: IV Placebo, enoxaparin
Drug: Placebo — Administered per the protocol
  Arms: IV Placebo, SC REGN7508; IV Placebo, apixaban; IV Placebo, enoxaparin

SUMMARY:
This study is researching an experimental drug called REGN7508 (called "study drug"). The study is focused on adults undergoing elective, unilateral (one side) total knee replacement surgery.

The aim of the study is to see how effective the study drug is at preventing venous thromboembolism (VTE) and other related diseases after total knee replacement surgery.

The study is looking at several other research questions, including:

* What side effects may happen from taking the study drug
* How much study drug is in the blood at different times
* Whether the body makes antibodies against the study drug (which could make the study drug less effective or could lead to side effects)

ELIGIBILITY:
Key Inclusion Criteria:

1. Is undergoing a primary elective unilateral TKA
2. Is in good health based on laboratory safety testing as described in the protocol
3. Body weight ≤130 kg at screening visit as described in the protocol

Key Exclusion Criteria:

1. Any condition that, as assessed by the investigator, may confound the results of the study or pose an additional risk to the participant by study participation
2. History of bleeding in the 6 months prior to randomization requiring hospitalization or transfusion as described in the protocol
3. History of thromboembolic disease or thrombophilia
4. History of major surgery, including brain, spinal, or ocular, or major trauma within approximately the past 6 months prior to randomization
5. Has an estimated Glomerular Filtration Rate (GFR) of <30 mL/min/1.73 m2 at the screening visit as described in the protocol

Note: Other protocol-defined Inclusion/ Exclusion Criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2027-02-20 (Estimated); Study Completion 2027-05-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of the composite endpoint of asymptomatic or symptomatic Venous Thromboembolism (VTE) [including VTE-related death] | Through day 12 visit, approximately 14 days

SECONDARY OUTCOMES:
Incidence of confirmed symptomatic Deep Venous Thrombosis (DVT) | Through day 12 visit, approximately 14 days
Incidence of confirmed Pulmonary Embolism (PE) | Through day 12 visit, approximately 14 days
Incidence of VTE-related death | Through day 12 visit, approximately 14 days
Incidence of the composite endpoint of major and clinically relevant non-major (CRNM) bleeding | Through day 12 visit, approximately 14 days
Incidence of the composite endpoint of asymptomatic or symptomatic VTE (including VTE-related death) | Through day 12 visit, approximately 14 days
Incidence of minor bleeding | Through day 12 visit, approximately 14 days
Incidence of Treatment Emergent Adverse Events (TEAEs) | Approximately day 90
Incidence of Anti-Drug Antibodies (ADA) to REGN7508 | Approximately day 90
Titer of ADA to REGN7508 | Approximately day 90
Concentrations of REGN7508 | Approximately day 90

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (33):
- United States (15):
  - Shoals Medical Trials, Inc., Sheffield, Alabama
  - CARI Clinical Trials, Riverside, California
  - Denver Metro Orthopedics, P.C. Englewood Location, Englewood, Colorado
  - Delray Physician Care Center, Delray Beach, Florida
  - Bioresearch Partner, Miami, Florida
  - Sacred Heart Health System Inc, Pensacola, Florida
  - Gulfcoast Research Institute, Sarasota, Florida
  - Phoenix Clinical Research, Tamarac, Florida
  - Sinai Hospital of Baltimore, Inc., Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Curalta Clinical Trials, Westwood, New Jersey
  - HD Research - First Surgical Hospital, Bellaire, Texas
  - NextStage Clinical Research, All American Orthopedics and Sports Medicine, Houston, Texas
  - Futuro Clinical Trials, McAllen, Texas
  - Flourish Research - San Antonio (Formerly Clinical Trials of Texas), San Antonio, Texas
- Bulgaria (2):
  - Multi-profile Hospital for Active Treatment Hearth and Brain EAD, Pleven
  - University Multiprofile Hospital for Active Treatment "Prof. Dr. Stoyan Kirkovich", Stara Zagora
- Semmelweis University, Budapest, Hungary
- Japan (6):
  - Kansai Rosai Hospital, Amagasaki-shi, Hyōgo
  - Yuuai Medical Center, Tomigusuku, Okinawa
  - National Hospital Organization Osaka Minami Medical Center, Kawachi-Nagano, Osaka
  - Osaka Saiseikai Nakatsu Hospital, Kita-Ku, Osaka
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Saga University Hospital, Saga
- Latvia (5):
  - Liepajas regionala slimnica; SIA, Liepāja
  - Rigas 2 slimnica, SIA, Riga
  - Hospital of Traumatology and Orthopaedics, Riga
  - ORTO Klinika, Riga
  - Vidzemes slimnica, Valmiera
- Lithuania (3):
  - Lietuvos sveikatos mokslu universiteto Kauno ligonine, Kaunas
  - Lietuvos sveikatos mokslu universiteto ligonine Kauno klinik, Kaunas
  - Vsi Klaipedos Universitetine Ligonine, Klaipėda
- Szpital Specjalistyczny im. Ludwika Rydygiera w Krakowie sp. z o.o., Krakow, Poland

IPD SHARING:
Plan to Share IPD: Yes
When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication, has made results publicly available (e.g., scientific publication, scientific conference, clinical trial registry), has the legal authority to share the data, and has ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/